CLINICAL TRIAL: NCT00675467
Title: Palliative Care and Symptom Management for the Pediatric Oncology Patient
Status: Completed | Type: Observational
Sponsor: M.D. Anderson Cancer Center (Other)
Responsible Party: Sponsor
Other Study IDs: 2007-0054
Record Dates: First submitted 2008-05-07; First posted 2008-05-09 (Estimated); Last update posted 2016-04-08 (Estimated); Status verified 2016-04

CONDITIONS: Pediatric Cancers
Keywords: Pediatric Cancer; Focus Group; Pediatric cancer patients; Parents of Pediatric cancer patients; Pediatric Palliative Care Program
MeSH Terms: conditions — Neoplasms | interventions — Caregivers

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (7):
- Group 1: Early cancer group-children ages 10-13 years
  Interventions: Behavioral: Focus Group - Parent/Caregiver; Behavioral: Focus Group - Pediatric Patient
- Group 2: Early cancer group-children ages 14 to 18 years
  Interventions: Behavioral: Focus Group - Parent/Caregiver; Behavioral: Focus Group - Pediatric Patient
- Group 3: Early cancer group-parents of patients ages 10-18 years
  Interventions: Behavioral: Focus Group - Parent/Caregiver; Behavioral: Focus Group - Pediatric Patient
- Group 4: Advanced cancer group-children ages 10-13 years
  Interventions: Behavioral: Focus Group - Parent/Caregiver; Behavioral: Focus Group - Pediatric Patient
- Group 5: Advanced cancer group-children ages 14-18 years
  Interventions: Behavioral: Focus Group - Parent/Caregiver; Behavioral: Focus Group - Pediatric Patient
- Group 6: Advanced cancer group-parents of children ages 10-18 years
  Interventions: Behavioral: Focus Group - Parent/Caregiver; Behavioral: Focus Group - Pediatric Patient
- Group 7: End of life group - parents of children ages birth to 18 years of age at time of death
  Interventions: Behavioral: Focus Group - Parent/Caregiver; Behavioral: Focus Group - Pediatric Patient

INTERVENTIONS:
Behavioral: Focus Group - Parent/Caregiver — A 1 1/2 hour group session with other parents/caregivers.
Behavioral: Focus Group - Pediatric Patient — A 1 1/2 hour group session with other pediatric patients.

SUMMARY:
The goal of this study is to learn about the communication, decision-making, symptom management, emotional adjustment, and spiritual needs of parents and pediatric patients treated at the Children's Cancer Hospital at M. D. Anderson (MCACC).

Primary Objectives:

1. Determine the palliative care service needs of pediatric cancer patients and their parents, including communication, decision-making, symptom management, emotional and spiritual support when receiving treatment for early cancer, treatment for advanced disease, and treatment in the end-of-life period.
2. Identify intra-group differences in the categories listed in Objective 1 for pediatric cancer patients receiving treatment (a) for early cancer, (b) for advanced disease, and (c) at end-of-life.

Secondary Objectives:

1. Inform the development of a Pediatric Palliative Care Program at the Children's Cancer Hospital at The University of Texas M. D. Anderson Cancer Center (MCACC or MDACC) based on identified needs as determined by primary study aims 1 and 2.

DETAILED DESCRIPTION:
PARENT:

The Focus Group:

If you agree to take part in this study, you will attend a 1 1/2 hour group session with 3-9 other caregivers. The group will be led by a group leader and an assistant. The group leader will ask questions to the group about communication, decision-making, symptom management, emotional adjustment, and spirituality experiences and needs during your child's treatment. If you have a child who is also taking part in this study, you will meet separately from your child.

At the time of your arrival and before the beginning of the focus group session, you will be asked to complete a questionnaire. You will be asked about you and your child's age, sex, where you live, your religion (if any), your ethnicity and race, and if there are other children in the family. You will be asked about when you found out your child had cancer, the type of cancer, and when the cancer got worse or came back (if applicable). You will be asked whether others have shared parenting responsibilities, your education level, and if you work and what type of work you do. The questionnaire will take about 5 minutes to complete.

Audiotapes/Transcripts:

The assistant will take notes and the session will be recorded on an audiotape. All audiotapes will be stored in locked cabinets maintained by the study chair. The audiotapes will be destroyed once the study and analyses are complete.

The audiotape will be recorded onto paper "transcripts". The completed focus group transcriptions will be placed in a database secured with a password and identification protected. Transcribed results will have all identifiable markers removed and kept in the investigators' locked files. Only the researchers will be able to view the transcriptions.

Length of Study:

Your participation on this study is complete once you finish the group meeting.

PEDIATRIC PARTICIPANT:

The Focus Group:

If you agree to take part in this study, you will go to a 1 1/2 hour group session with 3-9 other patients. The group will be led by a group leader and an assistant. The group leader will ask questions to the group about who you talk with about the disease, how you make a decision, how you manage any symptoms you may have, how you are feeling about the disease, and how religion has helped you during your treatment. If your parent is also taking part in this study, you will meet separately from your parent.

At the time of your arrival and before the beginning of the focus group session, your parent will be asked to complete a questionnaire. Your parent will be asked about their age and sex, your age and sex, where you live, your religion (if any), your ethnicity and race, and if there are other children in the family. Your parent will be asked when they found out you had cancer, the type of cancer, and when the cancer got worse or came back (if applicable). Your parent will be asked whether others have shared parenting responsibilities, their education level, and if they work and about the type of work they do. The questionnaire will take about 5 minutes to complete.

Audiotapes/Transcripts:

The assistant will take notes and the session will be recorded on an audiotape. All audiotapes will be stored in locked cabinets taken care of by the study chair. The audiotapes will be destroyed once the study is over and the researchers have finished looking at the information.

The audiotape will be recorded onto paper "transcripts". The completed focus group transcriptions will be placed in a database secured with a password and identification protected. Any personal information about you will be removed from these papers and the papers will be kept in the investigators' locked files. Only the researchers will be able to view the transcriptions.

Length of Study:

Your participation on this study is over once you complete the focus group.

ELIGIBILITY:
Inclusion Criteria:

Inclusion for Children:

* 10-18 years of age
* MD Anderson Children's Cancer Center (MCACC) cancer patient
* receiving anti-cancer treatment for disease that is not recurrent or metastatic for cancer diagnosed in the past 3-12 mos or receiving anti-cancer treatment for recurrent or metastatic cancer diagnosed within the past 3-12 months
* speak & understand English
* reside in the Greater Houston area
* provide IRB-approved pediatric assent or informed consent, as age appropriate
* if < 18 years of age, provide Internal Review Board (IRB)-approved parental permission
* child's eligibility is not contingent upon parent's decision to participate

Inclusion for parents:

* self-identified parent(s) that has(have) a child eligible for study, per the inclusion and exclusion criteria noted above or has had a child (0-18 yrs of age at time of death) treated for cancer at MCACC who has died in the last 1 to 2 years
* speak and understand English
* reside in the Houston metropolitan area
* provide IRB-approved informed consent
* attend different focus groups if more than one eligible parent per child (max 2 parents per child)
* parent's eligibility is not contingent upon the child's decision to participate

Exclusion Criteria:

Exclusion for Children:

* have cognitive impairment, developmental delay, or emotional distress that would limit participation in a group discussion, as determined by the clinical judgment of the investigator
* younger than 10 years or older than 18 years of age

Exclusion for Caregiver:

* have cognitive impairment, developmental delay, or emotional distress that would limit participation in a group discussion, as determined by the clinical judgment of the investigator.

Ages: 10 Years to 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Study Population: Study participants 10-18 years of age with cancer and their parent(s) or caregiver(s).
Sampling Method: Probability Sample
Enrollment: 13 (Actual)
Dates: Start 2008-04; Primary Completion 2016-04 (Actual)

PRIMARY OUTCOMES:
Palliative Care Service Needs of Pediatric Cancer Patients + Their Parents | 3 Years
  Qualitative data collection.

CONTACTS AND LOCATIONS:
Overall Officials: Rhonda Robert, PhD, Principal Investigator — M.D. Anderson Cancer Center
Locations (1):
- University of Texas MD Anderson Cancer Center, Houston, Texas, United States

REFERENCES:
- See also: University of Texas MD Anderson Cancer Center Website — http://www.mdanderson.org